CLINICAL TRIAL: NCT03373955
Title: A Prospective Study of Constructing Immune Repertoire Using Next-generation Sequencing (NGS) to Monitor the Therapeutic Effect in NSCLC Patients
Brief Title: A Prospective Study of Constructing Immune Repertoire to Monitor the Therapeutic Effect in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Oncology, Sichuan University
Other Study IDs: GHR-001
Record Dates: First submitted 2017-11-23; First posted 2017-12-14 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: T Cell repertoire; lung cancer; tumor mutation burden; Circulating tumour DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the investigators will extract Genomic DNA from peripheral blood and extract CtDNA from plasma ASAP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunotherapy,chemotherapy,radiotherapy: Pembrolizumab will be administered via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent.The peripheral blood will be collected at 3 weeks,2 months, 6 months,an average of 1 year
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — anti-programmed death 1 (PD-1) antibody

SUMMARY:
This study is designed to evaluate the untreated NSCLC patients. After participants have accepted chemotherapy, radiotherapy, and immunotherapy, the investigators used the next generation sequence technology (NGS) to construct immune repertoire to detective variation of patients' immune state and to monitor patients' therapeutic effect. The investigators are aim to explore the novel clone sequence as potential therapy target.

DETAILED DESCRIPTION:
Lung cancer was one of the most deadly tumors in the world. The standard of care for patients is platinum-based doublet chemotherapy concurrent with radiotherapy. As for patients with a mutant epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase(ALK), EGFR or ALK tyrosine kinase inhibitors (TKIs) are the standard first-line therapy. Now, the Food and Drug Administration approved Ipilimumab, Nivolumab, and Pembrolizumab as first-line or second-line therapy for NSCLC. However, there was no reports about therapeutic effect for NSCLC patients through detecting herself immune state, immune repertoire could explore patients' immune clonality and diversity using NGS technology.The investigators look forward to illuminate the mechanism of patients antitumor action.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified stage IV non-small cell lung cancer without treated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Pathology is mixed type•
* Poor vasculature
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of locally advanced or metastatic non small cell lung cancer progressed without previous treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
T cell repertoire | baseline, 2 months, 6 months, 1 year
  peripheral blood was collected at baseline,3 weeks,2 months, 6 months,an average of 1 year

SECONDARY OUTCOMES:
peripheral blood circulating tumor DNA | baseline, 2 months, 6 months, 1 year
  peripheral blood was collected at baseline,3 weeks,2 months, 6 months,an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Result] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Result] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Result] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Result] Yarchoan M, Johnson BA 3rd, Lutz ER, Laheru DA, Jaffee EM. Targeting neoantigens to augment antitumour immunity. Nat Rev Cancer. 2017 Apr;17(4):209-222. doi: 10.1038/nrc.2016.154. Epub 2017 Feb 24. PMID 28233802
- [Result] Ott PA, Hu Z, Keskin DB, Shukla SA, Sun J, Bozym DJ, Zhang W, Luoma A, Giobbie-Hurder A, Peter L, Chen C, Olive O, Carter TA, Li S, Lieb DJ, Eisenhaure T, Gjini E, Stevens J, Lane WJ, Javeri I, Nellaiappan K, Salazar AM, Daley H, Seaman M, Buchbinder EI, Yoon CH, Harden M, Lennon N, Gabriel S, Rodig SJ, Barouch DH, Aster JC, Getz G, Wucherpfennig K, Neuberg D, Ritz J, Lander ES, Fritsch EF, Hacohen N, Wu CJ. An immunogenic personal neoantigen vaccine for patients with melanoma. Nature. 2017 Jul 13;547(7662):217-221. doi: 10.1038/nature22991. Epub 2017 Jul 5. PMID 28678778
- [Result] Khodadoust MS, Olsson N, Wagar LE, Haabeth OA, Chen B, Swaminathan K, Rawson K, Liu CL, Steiner D, Lund P, Rao S, Zhang L, Marceau C, Stehr H, Newman AM, Czerwinski DK, Carlton VE, Moorhead M, Faham M, Kohrt HE, Carette J, Green MR, Davis MM, Levy R, Elias JE, Alizadeh AA. Antigen presentation profiling reveals recognition of lymphoma immunoglobulin neoantigens. Nature. 2017 Mar 30;543(7647):723-727. doi: 10.1038/nature21433. Epub 2017 Mar 22. PMID 28329770
- [Result] Robbins PF, Kassim SH, Tran TL, Crystal JS, Morgan RA, Feldman SA, Yang JC, Dudley ME, Wunderlich JR, Sherry RM, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Li YF, El-Gamil M, Rosenberg SA. A pilot trial using lymphocytes genetically engineered with an NY-ESO-1-reactive T-cell receptor: long-term follow-up and correlates with response. Clin Cancer Res. 2015 Mar 1;21(5):1019-27. doi: 10.1158/1078-0432.CCR-14-2708. Epub 2014 Dec 23. PMID 25538264
- [Result] Apetoh L, Ghiringhelli F, Tesniere A, Obeid M, Ortiz C, Criollo A, Mignot G, Maiuri MC, Ullrich E, Saulnier P, Yang H, Amigorena S, Ryffel B, Barrat FJ, Saftig P, Levi F, Lidereau R, Nogues C, Mira JP, Chompret A, Joulin V, Clavel-Chapelon F, Bourhis J, Andre F, Delaloge S, Tursz T, Kroemer G, Zitvogel L. Toll-like receptor 4-dependent contribution of the immune system to anticancer chemotherapy and radiotherapy. Nat Med. 2007 Sep;13(9):1050-9. doi: 10.1038/nm1622. Epub 2007 Aug 19. PMID 17704786
- [Result] Herrera FG, Bourhis J, Coukos G. Radiotherapy combination opportunities leveraging immunity for the next oncology practice. CA Cancer J Clin. 2017 Jan;67(1):65-85. doi: 10.3322/caac.21358. Epub 2016 Aug 29. PMID 27570942
- [Result] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329